CLINICAL TRIAL: NCT05625828
Title: Evaluation of the Effects of a Cognitive-Motor Fall Prevention Program "SILVER XIII - EQUILIBRE" on Fall Risk Factors: Functional Abilities and Executive Functions
Brief Title: Evaluation of the Effects of a Cognitive-Motor Fall Prevention Program on Fall Risk Factors
Acronym: 13EVAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EZUS-LYON 1 (Other)
Collaborators: Laboratoire Interuniversitaire de Biologie de la Motricité (Other); Centre Hospitalier de Roanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 005B2022
Record Dates: First submitted 2022-11-04; First posted 2022-11-23 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Accidental Falls; Aging; Mild Cognitive Impairment
Keywords: Dual-Task; Physical Activity; Prevention
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SILVER XIII EQUILIBRE (Experimental): Cognitive-motor 10 weeks program
  Interventions: Behavioral: Cognitive-motor Physical Activity
- VIVIFRAIL (Active Comparator): Multifactorial 10 weeks program
  Interventions: Behavioral: Multifactorial Physical Activity

INTERVENTIONS:
Behavioral: Cognitive-motor Physical Activity — Physical activity program that consist of 1 sessions per week during 10 weeks (from Week 2 to Week 11). Each session includes a 10 minutes warm up with light walking, 45 minutes of cognitive-motor exercises where participants have to perform two tasks consequently (for example, walking while answering math questions or throwing a ball while reverse walking) and 5 minutes of stretching exercises.
  Arms: SILVER XIII EQUILIBRE
Behavioral: Multifactorial Physical Activity — Physical activity program that consist of 1 sessions per week during 10 weeks (from Week 2 to Week 11). Each session includes a 10 minutes warm up with light walking, 45 minutes of multifactorial exercises that consists of high speed walking, resistance training and balance training in single task condition and 5 minutes of stretching exercises.
  Arms: VIVIFRAIL

SUMMARY:
The goal of this interventional study is to compare in community dwelling elderly people the effects of two physical activity programs to prevent accident falls : "SILVER XIII EQUILIBRE" program and "VIVIFRAIL" program, on several risks factors such as executive functions and functional capacities.

Participants will perform a 1 hour physical activity session during 10 weeks and effects will be measured using a multidimensional test battery. "SILVER XIII EQUILIBRE" program contains cognitive-motor exercises where participants have to perform two tasks simultaneously such as answering math questions while walking whereas "VIVIFRAIL" program contains multifactorial exercises such as walking, balance training and resistance training in single-task condition.

The main question it aims to answer is :

• Does physical activity enriched with simultaneous cognitive exercises enhances the effects ?

DETAILED DESCRIPTION:
Falls in the elderly are a problem of increasing importance in our aging societies. Among the multiple intrinsic risk factors, if the age-induced decline of functional and locomotor capacities are recognized risk factors, impaired executive functioning is another equally important one. Thus, Mild Cognitive Impairment (MCI) - characterized by an early deficit in executive functioning but not pathological - turns out to be an independent and significant risk factor. In order to reduce the impact of this problem and thus promote "well aging", it is essential to develop effective preventive approaches on all of these risk factors. Of these, cognitive-motor fall prevention programs - based on simultaneous cognitive and motor tasks - are the most effective in reducing the rate of falls. However, since 2017, the French Rugby League Federation has been proposing such an innovative program called "SILVER XIII - EQUILIBRE" consisting of 10 one-hour sessions per week and including a majority of cognitive-motor exercises. In addition, this program also includes exercises for learning the "play the ball", a specific skill of rugby league that consist of shooting the ball with the heel and making a step forward which is close to the stepping strategy to avoid falling. Initially intended for community dwelling elderly people and non-fallers presenting a usual aging (average age = 67.6 +/- 3 years), it turns out that this program welcomes three different profiles of elderly people that we find in the literature: (1) young-aged, active people with no deficits in functional and cognitive abilities; (2) older people with optimal cognitive aging but less active (3) older people with MCI. As the effects of regular Physical Activity (PA) depend on the initial level of each individual, it could be that the effects of the "SILVER XIII - EQUILIBRE" program on both functional abilities and executive functions depend on the profile of the elderly. In order to answer the main question the effects of the "SILVER XIII EQUILIBRE" program will be compared to an active comparator : the "VIVIFRAIL" program which is a international multifactorial program to prevent falls based on walking, balance and resistance training single task exercises.

ELIGIBILITY:
Inclusion Criteria:

* Older people living at home
* Able to walk without technical assistance

Exclusion Criteria:

* Presence of a proven major neurocognitive disorder (MOCA score < 18)
* Patients with severe depression (Geriatric Depression Scale score > 10)
* Body mass index (BMI) > 35
* Diagnosed and known neurological or neurodegenerative pathology
* Having declared more than 3 falls in the pas year
* Presence of a motor disorder
* Contraindication to the practice of a physical or sporting activity
* Participation in another protocol for the prevention of falls or loss of autonomy in the last 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 176 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-10-24 (Estimated)

PRIMARY OUTCOMES:
Change of Trail Making Test part A and B scores at Week 12 after intervention | Week 1 and Week 12
  Participants will be asked to perform the Trail Making Test part A and B (Reitan, 1958) following the instructions of the evaluator. It consist of connecting by making pencil lines 25 encircled numbers randomly arranged on a page in proper order (part A) and 25 encircled numbers and letters in alternating order (part B). A sample page including only 8 circles is made for training just before each 25 circle test page. Measurements will take place one week before the first session (Week 1) and one week after the last session (Week 12). Execution time will be measured in seconds.
Change of Stroop Test Victoria version scores at Week 12 after intervention | Week 1 and Week 12
  Participants will be asked to perform the Stroop Test Victoria version (Bayard, 2011) following the instructions of the evaluator. It consist of three pages each containing 6 lines of 4 items and each page includes an additional line for training. In the page 1 participant has to tell the color of 4 dots printed in color ink in left to right order and line by line ; in the page two 4 neutral words are printed in color ink and participants has to tell the color of the ink in the same order ; in page three 4 color words are printed in color ink and participants has to tell the color of the ink in the same order. Measurements will take place one week before the first session (Week 1) and one week after the last session (Week 12). Execution time in second and errors will be measured.
Change of walking speed at Week 12 after intervention | Week 1 and Week 12
  Participants will perform a 6 meters gait measurement where they have to walk at self pace on a 10 meters corridor and time in second will be measured on 6 meters using photoelectric sensors. The first 2 meters are for reaching the pace and last 2 meters are to stop. Measurements will take place one week before the first session (Week 1) and one week after the last session (Week 12). Spontaneous gait speed will be measured in meters per second.

SECONDARY OUTCOMES:
Change of Choice Stepping Reaction Time at Week 12 after intervention | Week 1 and Week 12
  Participants will perform a Choice Stepping Reaction Task (Lord SR & Fitzpatrick, 2001) : Participants stand on a nonslip black platform that contained four rectangular panels, one in the front one in the back and one to the side of each foot (up, down, left and right). A computer generates a stimuli (an arrow) indicating the direction of the target the participant has to step on as fast as possible. Choice Stepping Reaction Time that consist of time between the presentation of stimuli and the foot lift will be measured in second. Measurements will take place one week before the first session (Week 1) and one week after the last session (Week 12).
Change of 30 second sit to stand test score at Week 12 after intervention | Week 1 and Week 12
  This test is a part of the Senior Fitness Test assessment (Fournier et al., 2012). Participants will perform the 30 second sit to stand test, which consist of repetitively standing up from a chair as fast as possible during 30 seconds. Measurements will take place one week before the first session (Week 1) and one week after the last session (Week 12). Number of repetition will be measured.
Change of 2 minutes step in place test at Week 12 after intervention | Week 1 and Week 12
  This test is a part of the Senior Fitness Test assessment (Fournier et al., 2012). Participants will perform the 2 minutes step in place test which consist of alternatively lifting the knees to an height given by the evaluator as fast as possible during 2 minutes. Measurements will take place one week before the first session (Week 1) and one week after the last session (Week 12). Number of repetitions (corresponding of each knee lift) will be measured.
Change of one leg standing position time at Week 12 after intervention | Week 1 and Week 12
  This test is a part of the Senior Fitness Test assessment (Fournier et al., 2012). Participants will be asked to stay on one leg standing position and the maximal time they managed to maintain the position will be measured in seconds. Measurements will take place one week before the first session (Week 1) and one week after the last session (Week 12).
Change of dual-task walking speed at Week 12 after intervention | Week 1 and Week 12
  Participants will perform a 6 meters gait measurement where they have to walk at self pace on a 10 meters corridor and time in second will be measured on 6 meters using photoelectric sensors. The first 2 meters are for reaching the pace and last 2 meters are to stop. Participants have to walk doing the following cognitive tasks. An arithmetic task : Participants have to continuously substract 7 to a 3 digit number given by the evaluator giving results orally. Percentage of error in the cognitive task will be measured and spontaneous gait speed in meters per second will be measured. Measurements will take place one week before the first session (Week 1) and one week after the last session (Week 12).
Change in the walking trail making test outcomes at Week 12 after intervention | Week 1 and Week 12
  Participants will perform the "Walking Trail Making Test" (WTMT) Task (Alexander et al., 2005 ; Perrochon et al., 2014) on a 10 meters corridor and time in second will be measured on 6 meters using photoelectric sensors. The first 2 meters are for reaching the pace and last 2 meters are to stop. The WTMT contains three experimental conditions : WTMT-N in which participants have to step on numbers from 1 to 20 in ascending order ; WTMT-A in which participants have to step on the same numbers avoiding numeric distractors ; WTMT-B in which participants have to step alternatively on numbers and letters following ascending order and alphabetic order avoiding numeric and alphabetic distractors. Percentage of error and execution time in seconds will be measured. Measurements will take place one week before the first session (Week 1) and one week after the last session (Week 12)
Change in fall rate at Week 36 after intervention | From Week 12 to Week 36
  Fall rate will be measured using a 6 month follow up. Participants will be asked to fill in an online weekly report indicates whether they had falls or not during the past week.
Global cognition score at Week 1 | Week 1
  Participants will be asked to perform the different steps of the Montreal Cognitive Assessment following the instructions of the evaluator. This test evaluates multiple cognitive functions such as executive functions, memory, attention leading to a score between 0 (worse score) and 30 (best score). A score between 0 and 20 indicates a major cognitive impairment, a score between 20 and 25 indicates a mild cognitive impairment and and score superior to 25 indicates normal cognitive functioning. Measurement will take place one week before the first session (Week 1).
Fall Risk score at Week 1 | Week 1
  Fall Risk will be measured using a 7 items questionnaire (Bongue et al., 2011) leading to a score between 0 (best score) and 12 (worst score). A score between 0 and 3 indicates a low risk of falling, a score between 4 and 7 indicates a moderate risk of falling and a score superior to 7 indicates a high risk of falling. Measurements will take place one week before the first session (Week 1).
Common physical activity at Week 1 | Week 1
  Using a self-reported questionnaire named "Physical Activity Questionnaire for the Elderly ", participants will be asked to register all the physical activities they had on the past week and the time allowed to each activity (De Souto-Barretto et al., 2011). The amount of physical activity will be measured in Metabolic Equivalent Task per minutes per week. Measurements will take place one week before the first session (Week 1).
Sedentary behaviors at Week 1 | Week 1
  Using a self-reported questionnaire named "Recent Physical Activity Questionnaire" (Golubic et al., 2014), participants will be asked to register all the sedentary behaviors they have usually each day and the time allowed to each behavior. The amount sedentary behavior will be measured in hour per day. Measurements will take place one week before the first session (Week 1).

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Fabre, MD, Study Director — Centre Hospitalier de Roanne; Pascal Chabaud, PhD, Study Director — Laboratoire Inter-universitaire de Biologie de la Motricité, UR7424; Rafael Mauti, MSc, Principal Investigator — Laboratoire Inter-universitaire de Biologie de la motricité, UR7424
Locations (1):
- Laboratoire Inter-universitaire de Biologie de la Motricité, UR7424, Villeurbanne, Rhône, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayard S, Erkes J, Moroni C; College des Psychologues Cliniciens specialises en Neuropsychologie du Languedoc Roussillon (CPCN Languedoc Roussillon). Victoria Stroop Test: normative data in a sample group of older people and the study of their clinical applications in the assessment of inhibition in Alzheimer's disease. Arch Clin Neuropsychol. 2011 Nov;26(7):653-61. doi: 10.1093/arclin/acr053. Epub 2011 Aug 26. PMID 21873625
- [Background] REITAN RM. The relation of the trail making test to organic brain damage. J Consult Psychol. 1955 Oct;19(5):393-4. doi: 10.1037/h0044509. No abstract available. PMID 13263471
- [Background] Lord SR, Fitzpatrick RC. Choice stepping reaction time: a composite measure of falls risk in older people. J Gerontol A Biol Sci Med Sci. 2001 Oct;56(10):M627-32. doi: 10.1093/gerona/56.10.m627. PMID 11584035
- [Background] Bongue B, Dupre C, Beauchet O, Rossat A, Fantino B, Colvez A. A screening tool with five risk factors was developed for fall-risk prediction in community-dwelling elderly. J Clin Epidemiol. 2011 Oct;64(10):1152-60. doi: 10.1016/j.jclinepi.2010.12.014. Epub 2011 Apr 3. PMID 21463927
- [Background] Fournier J, Vuillemin A, Le Cren F. Mesure de la condition physique chez les personnes âgées. Evaluation de la condition physique des seniors : adaptation française de la batterie américaine " Senior Fitness Test ". Science & Sport. 2012; 27 : 254-259.
- [Background] De Souto Barreto, P., Ferrandez, A. M., & Saliba-Serre, B. Questionnaire d'activité physique pour les personnes âgées (QAPPA): validation d'un nouvel instrument de mesure en langue française. Science and Sports. 2011; 26(1): 11-18.
- [Background] Golubic R, May AM, Benjaminsen Borch K, Overvad K, Charles MA, Diaz MJ, Amiano P, Palli D, Valanou E, Vigl M, Franks PW, Wareham N, Ekelund U, Brage S. Validity of electronically administered Recent Physical Activity Questionnaire (RPAQ) in ten European countries. PLoS One. 2014 Mar 25;9(3):e92829. doi: 10.1371/journal.pone.0092829. eCollection 2014. PMID 24667343
- [Background] Perrochon A, Kemoun G. The Walking Trail-Making Test is an early detection tool for mild cognitive impairment. Clin Interv Aging. 2014;9:111-9. doi: 10.2147/CIA.S53645. Epub 2014 Jan 7. PMID 24426778
- [Background] Alexander NB, Ashton-Miller JA, Giordani B, Guire K, Schultz AB. Age differences in timed accurate stepping with increasing cognitive and visual demand: a walking trail making test. J Gerontol A Biol Sci Med Sci. 2005 Dec;60(12):1558-62. doi: 10.1093/gerona/60.12.1558. PMID 16424288